CLINICAL TRIAL: NCT05043844
Title: Effect of Abdominal Binder Use on Postoperative Shoulder Pain After Laparoscopic Gynecological Surgery
Brief Title: Comparison of the Incidence of Shoulder Pain According to Postoperative Use of Abdominal Binder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2107-220-1240
Record Dates: First submitted 2021-08-27; First posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Shoulder Pain
Keywords: Laparoscopic Surgery; Gynecology
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): In the control group, an investigator performed only a pulmonary recruitment maneuver on the Trendelenburg position before the emergence of anesthesia.
- Abdominal binder (Experimental): In the abdominal binder group, a pulmonary recruitment maneuver was performed on the Trendelenburg position and the abdominal binder which had a standard height of 22 cm was placed on the abdomen of the patient before the emergence of anesthesia.
  Interventions: Device: abdominal binder

INTERVENTIONS:
Device: abdominal binder — Wearing an abdominal binder postoperatively
  Arms: Abdominal binder

SUMMARY:
The aim of the study is to evaluate the effect of the use of an abdominal binder on postoperative shoulder pain according to laparoscopic gynecological surgery. The investigators will compare the incidences of shoulder pain after laparoscopic gynecological surgery in terms of the use of an abdominal binder.

DETAILED DESCRIPTION:
Laparoscopic surgery has advantages over laparotomy in that it reduces postoperative pain and hospital stay. However, postoperative shoulder pain is one of the major concerns of laparoscopic surgery. Shoulder pain has been reported to occur in 35 to 70% of laparoscopic surgeries. The exact mechanism of shoulder pain after laparoscopic surgery is not clear. The main hypothesis is that the presence of residual carbon dioxide (CO2) in the abdominal cavity stimulates the diaphragmatic nerve and causes pain in the shoulder. Alveolar recruitment maneuver in the Trendelenburg position reduced the intensity and incidence of shoulder pain significantly. However, even with these measures, shoulder pain occurred in 63% of patients after surgery. In addition to this measure, The investigators hypothesized that wearing an abdominal binder would promote the absorption of residual CO2 in the abdominal cavity into the peritoneum and pelvis pressure.

The aim of this study was to evaluate the effect of the use of an abdominal binder on shoulder pain after gynecological laparoscopic surgery.

The intraoperative management is carried out in the same manner, except for wearing an abdominal binder after surgery. Laparoscopic procedure is completed, and then intraperitoneal CO2 is passive drained. An anesthetist places the operating table in the Trendelenburg position at 30 degrees and performs the alveolar recruitment maneuver. (CPAP 45 cm H2O is administered 5 times for 7 seconds) In the abdominal binder group, the patient wears an abdominal binder in the Trendelenburg position and then changed to the supine position before the emergence.

In the control group, the patient placed in the supine position, and emergence is started.

Shoulder pain at 12, 24, and 36 hours after surgery is investigated with a Numeric Score Scale (NRS) score.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 20-79 years with ASA I - III undergoing elective laparoscopic gynecological surgery under general anesthesia

Exclusion Criteria:

* Patients who do not consent to the trial
* Conversion to open surgery from laparoscopic surgery
* Patients with previous shoulder disease or history of shoulder surgery
* Patients who have difficulty wearing an abdominal binder due to skin disease or wounds in the abdomen
* Development of subcutaneous emphysema
* Change of intra-abdominal carbon dioxide pressure due to surgical difficulties

Ages: 20 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Postoperative shoulder pain | Postoperative shoulder pain at 12 hours after surgery
  Investigate occurrence of postoperative shoulder pain at 12 hours, 24 hours, and 36 hours after surgery. The occurrence of shoulder pain is defined as having NRS ≥ 1 pain at least once out of the three measurement time points.
Postoperative shoulder pain | Postoperative shoulder pain at 24 hours after surgery
  Investigate occurrence of postoperative shoulder pain at 12 hours, 24 hours, and 36 hours after surgery. The occurrence of shoulder pain is defined as having NRS ≥ 1 pain at least once out of the three measurement time points.
Postoperative shoulder pain | Postoperative shoulder pain at 36 hours after surgery
  Investigate occurrence of postoperative shoulder pain at 12 hours, 24 hours, and 36 hours after surgery. The occurrence of shoulder pain is defined as having NRS ≥ 1 pain at least once out of the three measurement time points.

SECONDARY OUTCOMES:
Intensity of postoperative shoulder pain | at 12 hours, 24 hours, and 36 hours after surgery
  Investigate shoulder pain intensity using numerical rating scale (0-10, 0 representing 'no pain', 10 representing 'worst pain imaginable')
Shoulder pain depending on posture | at 12 hours, 24 hours, and 36 hours after surgery
  Investigate whether there is a change in shoulder pain depending on the posture.
Surgical site pain | at 12 hours, 24 hours, and 36 hours after surgery
  Investigate Intensity of surgical site pain using numerical rating scale (0-10, 0 representing 'no pain', 10 representing 'worst pain imaginable')
Incidence of postoperative nausea and vomiting (PONV) | at 12 hours, 24 hours, and 36 hours after surgery
  The occurrence of PONV is defined as having PONV at least once out of the three measurement time points.
Time of first walking postoperatively | After transfer to general ward up to 36 hours
  Time of first walking after transfer to general ward

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, M.D., PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dobbs FF, Kumar V, Alexander JI, Hull MG. Pain after laparoscopy related to posture and ring versus clip sterilization. Br J Obstet Gynaecol. 1987 Mar;94(3):262-6. doi: 10.1111/j.1471-0528.1987.tb02365.x. PMID 2952160
- [Background] Ko-Iam W, Paiboonworachat S, Pongchairerks P, Junrungsee S, Sandhu T. Combination of etoricoxib and low-pressure pneumoperitoneum versus standard treatment for the management of pain after laparoscopic cholecystectomy: a randomized controlled trial. Surg Endosc. 2016 Nov;30(11):4800-4808. doi: 10.1007/s00464-016-4810-4. Epub 2016 Feb 23. PMID 26905574
- [Background] Phelps P, Cakmakkaya OS, Apfel CC, Radke OC. A simple clinical maneuver to reduce laparoscopy-induced shoulder pain: a randomized controlled trial. Obstet Gynecol. 2008 May;111(5):1155-60. doi: 10.1097/AOG.0b013e31816e34b4. PMID 18448749
- [Background] Korell M, Schmaus F, Strowitzki T, Schneeweiss SG, Hepp H. Pain intensity following laparoscopy. Surg Laparosc Endosc. 1996 Oct;6(5):375-9. PMID 8890423
- [Background] Sarli L, Costi R, Sansebastiano G, Trivelli M, Roncoroni L. Prospective randomized trial of low-pressure pneumoperitoneum for reduction of shoulder-tip pain following laparoscopy. Br J Surg. 2000 Sep;87(9):1161-5. doi: 10.1046/j.1365-2168.2000.01507.x. PMID 10971421
- [Background] Esmat ME, Elsebae MM, Nasr MM, Elsebaie SB. Combined low pressure pneumoperitoneum and intraperitoneal infusion of normal saline for reducing shoulder tip pain following laparoscopic cholecystectomy. World J Surg. 2006 Nov;30(11):1969-73. doi: 10.1007/s00268-005-0752-z. PMID 17043939
- [Background] Tsai HW, Chen YJ, Ho CM, Hseu SS, Chao KC, Tsai SK, Wang PH. Maneuvers to decrease laparoscopy-induced shoulder and upper abdominal pain: a randomized controlled study. Arch Surg. 2011 Dec;146(12):1360-6. doi: 10.1001/archsurg.2011.597. PMID 22184293
- [Background] Berberoglu M, Dilek ON, Ercan F, Kati I, Ozmen M. The effect of CO2 insufflation rate on the postlaparoscopic shoulder pain. J Laparoendosc Adv Surg Tech A. 1998 Oct;8(5):273-7. doi: 10.1089/lap.1998.8.273. PMID 9820719
- [Background] Das K, Karateke F, Menekse E, Ozdogan M, Aziret M, Erdem H, Cetinkunar S, Ozdogan H, Sozen S. Minimizing shoulder pain following laparoscopic cholecystectomy: a prospective, randomized, controlled trial. J Laparoendosc Adv Surg Tech A. 2013 Mar;23(3):179-82. doi: 10.1089/lap.2012.0410. Epub 2012 Dec 20. PMID 23256585
- [Background] Zeeni C, Chamsy D, Khalil A, Abu Musa A, Al Hassanieh M, Shebbo F, Nassif J. Effect of postoperative Trendelenburg position on shoulder pain after gynecological laparoscopic procedures: a randomized clinical trial. BMC Anesthesiol. 2020 Jan 29;20(1):27. doi: 10.1186/s12871-020-0946-9. PMID 31996139
- [Background] Kimura Kuroiwa K, Shiko Y, Kawasaki Y, Aoki Y, Nishizawa M, Ide S, Miura K, Kobayashi N, Sehmbi H. Phrenic Nerve Block at the Azygos Vein Level Versus Sham Block for Ipsilateral Shoulder Pain After Video-Assisted Thoracoscopic Surgery: A Randomized Controlled Trial. Anesth Analg. 2021 Jun 1;132(6):1594-1602. doi: 10.1213/ANE.0000000000005305. PMID 33332919